CLINICAL TRIAL: NCT00412776
Title: A Randomized, Multicentre Therapeutic Confirmatory Study to Evaluate the Efficacy and Safety of Proxinium Plus Best Supportive Care Versus Best Supportive Care Alone in Patients With Advanced SCCHN Who Have Received at Least One Anti-cancer Treatment Regimen for Advanced Disease
Brief Title: Study of Proxinium Plus Best Supportive Care Versus Best Supportive Care for Patients With Advanced Head and Neck Cancer
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Corporate reasons unrelated to safety and efficacy
Sponsor: Sesen Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VB4-845-01-IIIA
Record Dates: First submitted 2006-12-14; First posted 2006-12-18 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-12

CONDITIONS: Carcinoma, Squamous Cell of Head and Neck; Carcinoma, Squamous Cell; Neoplasms, Squamous Cell; Head and Neck Neoplasms; Mouth Neoplasms; Head and Neck Cancer
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Squamous Cell; Neoplasms, Squamous Cell; Head and Neck Neoplasms; Mouth Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Proxinium plus Best Supportive Care
  Interventions: Drug: Proxinium
- 2 (No Intervention): Best Supportive Care

INTERVENTIONS:
Drug: Proxinium — 700 µg Proxinium, once weekly until complete resolution of all target tumours or radiographic tumour progression
  Arms: 1

SUMMARY:
The purpose of this study is to compare the safety and efficacy of Proxinium plus best supportive care with best supportive care only for patients with squamous cell head and neck cancer.

DETAILED DESCRIPTION:
Head and neck cancer is a general description of a disease that includes several types of soft tissue carcinomas that develop in the head and neck regions.

Proxinium is a recombinant fusion protein that binds to the epithelial cell adhesion molecule (Ep-CAM) that is highly expressed on squamous cell carcinomas of the head and neck (SCCHN). Proxinium is administered via intratumoural injection.

The primary objective of the study is to compare the overall survival time for patients treated with intratumourally injected Proxinium plus BSC versus BSC alone. Secondary objectives of the study include comparison of locoregional tumour control, local progression-free survival, symptomatic benefit and safety profile in patients who receive Proxinium plus BSC versus patients who receive BSC

ELIGIBILITY:
Inclusion Criteria:

Disease Characteristics

* The patient must be 18 years of age or older.
* The patient must have squamous cell carcinoma of the head and neck.
* The squamous cell carcinoma must be Ep-CAM positive.
* ECOG performance status of 0, 1, 2 or 3.
* 12 week life expectancy

Prior/Concurrent Therapy

* The patient must have received therapy for their primary disease (eg, surgery and/or radiotherapy, chemo-radiotherapy or chemotherapy).
* The patient must have been diagnosed with persistent or recurrent disease or a second primary tumour.
* The patient's disease must be refractory.
* There must be at least 2 weeks between the last dose of chemotherapy or radiotherapy and receiving study drug or 4 weeks between the last dose of an experimental drug and receiving study drug.

Patient Characteristics

* The patient must have adequate hepatic function [alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 × upper limit of normal (ULN) and bilirubin level ≤1.5 × ULN].
* The patient must have adequate renal function (serum creatinine < 1.5 × ULN).
* The patient must have the following hematological values: granulocytes ≥1500/μL, platelets ≥75 000/μL and hemoglobin >8 g/dL.
* The patient must have prothrombin time and partial thromboplastin time within normal limits.

Other

• Women of childbearing potential and male patients must agree to use a highly effective contraceptive method.

Exclusion Criteria:

* The patient has clinically significant distant metastases.
* The patient is eligible to have surgical resection or radiotherapy, chemo-radiotherapy or chemotherapy.
* The patient has a nasopharyngeal tumour.
* The patient has AIDS, hepatitis C or hepatitis B.
* The patient has clinically significant renal or hepatic disease.
* Tumors are prone to bleeding.
* The patient is pregnant or lactating.
* The patient requires 'blood thinning' medications and can not safely discontinue the medication.
* The patient is currently enrolled in another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2005-12; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Survival | Death or 12 months from the date that the last patient required for efficacy analysis has been randomized

SECONDARY OUTCOMES:
Tumour response, safety and quality of life | Death or 12 months from the date that the last patient required for efficacy analysis has been randomized

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Cuthbert, Study Director — Viventia Biotech Inc.
Locations (122):
- Argentina (8):
  - Hospital Italiano Regional del Sur, Bahía Blanca
  - Hospital Municipal de Agudos Leonidas Lucero, Bahía Blanca
  - Centro de Estudio y Tratamiento de las Enfermedades Neoplasicas (CETEN), Buenos Aires
  - Hospital de Clinicas "Jose de San Martin", Buenos Aires
  - Hospital Nacional Alejandro Posadas, Buenos Aires
  - Hospital Universitario Austral, Buenos Aires
  - Instituto Medico Platense, La Plata
  - Hospital Italiano Garibaldi, Rosario
- Brazil (17):
  - Hospital de Câncer de Barretos - Fundação Pio XII, Barretos
  - Cettro - Centro de Tratamento Oncológico Ltda., Brasília
  - Centro Regional Integrado de Oncologia - CRIO, Fortaleza
  - Hospital Araújo Jorge, Goiania - GO
  - Hospital Amaral Carvalho, Jaú
  - Pro-Onco Centro De Tratamento Oncológico S/C Ltda, Londrina
  - Biocor - Hospital de Doenças Cardiovasculares Ltda, Nova Lima
  - CECAN - Centro do Câncer Francisco Cunha Filho, Piracicaba
  - Hospital São Lucas da PUCRS, Porto Alegre - RS
  - Irmandade Santa Casa de Misericórdia de Porto Alegre, Porto Alegre - RS
  - Instituto Ribeirãopretano de Combate ao Câncer, Riberao Preto-SP
  - INCA - Instituto Nacional do Câncer, Rio de Janeiro
  - SOS Vida - Soluções em Saúde, Salvador - BA
  - Santo André Diagnósticos e Tratamentos Ltda, Santo Andre-SP
  - Hospital Do Câncer A. C. Camargo, São Paulo
  - Grupo de Pesquisas Médicas, São Paulo - SP
  - Hospital das Clínicas - Faculdade de Medicina da Universidade de São Paulo, São Paulo - SP
- Croatia (3):
  - Clinical Hospital "Sestre milosrdnice", Zagreb
  - Clinical Hospital Centre Zagreb, Clinic for ENT, Department for Head and Neck Surgery, Zagreb
  - Universtity Hospital for Tumors, Department for Head and Neck Surgery, Zagreb
- France (3):
  - Centre Georges-Francois Leclerc, Dijon
  - Clinique Guillaume Le Conquerant, Le Havre
  - Centre Régional de Lutte contre le Cancer Val d'Aurelle, Montpellier
- Germany (9):
  - Charité -Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Köln, Cologne
  - Medizinische Hochschule Hannover, Hanover
  - Universität Heidelberg, Heidelberg
  - Universitätsklinikum Leipzig, Leipzig
  - Universitätsklinikum Schleswig Holstein, Lübeck
  - Johannes Gutenberg-Universität, Mainz
  - Klinikum der Philipps-Universität Marburg, Marburg
  - Universitätsklinikum Tübingen, Tübingen
- Hungary (4):
  - Fovarosi Onkormanyzat Uzsoki utcai Korhaza, Fej-nyaksebeszet, Budapest
  - Orszagos Onkologiai Intezet, Budapest
  - Debreceni Egyetem OEC, Onkologiai Tanszek, Debrecen
  - Petz Aladar Megyei Korhaz, Ful-orr-gege, Fej, Nyak Sebeszet, Győr
- India (17):
  - Department of Medical Oncology, Bangalore Institute of Oncology, Bangalore
  - Kidwai Memorial Institute of Oncology, Bangalore
  - Global Hospitals, Hyderabaad
  - MNJ Institute of Oncology, Hyderabaad
  - Nizam's Institute of Medical Sciences, Hyderabaad
  - Birla Cancer Institute SMS Medical College Hospital, Jaipur
  - SK Soni Hospital, Jaipur
  - Soumya Hospita, Karkhāna
  - Amrita Institute of Medical Sciences and Research Centre, Kochi
  - Netaji Subash Chandra Bose Cancer Research Institute, Kolkata
  - Orchid Nursing Home, Kolkata
  - Department of Medical Oncology Dayanand Medical College & Hospital, Ludhiana
  - Asian Institute of Oncology, S L Raheja Hospital, Mumbai
  - Tata Memorial Hospital, Mumbai
  - Department of Medical Oncology AIIMS, Institute Rotary Cancer Hospital, New Delhi
  - Department of Medical Oncology Rajiv Gandhi Cancer Institute and Research Centre, New Delhi
  - Regional Cancer Centre, Trivandrum
- Israel (7):
  - Soroka University Medical Center, Beersheba
  - The Lady Davis Carmel Medical Center, Haifa
  - Haddasa Ein Carem Hospital, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Kaplan Medical Center, Rehovot
  - Tel Aviv University Medical School, Tel Aviv
  - Sheba - Medical Center, Tel Litwinsky
- Italy (3):
  - Azienda Ospedaliera San Gerardo, Monza
  - IRCCS Policlinico San Matteo, Pavia
  - Azienda Ospedaliera Pisana, Pisa
- Mexico (5):
  - Hospital Clínica del Parque, Chihuahua, Chih.
  - Centro Anticanceroso de la Cruz Roja Mexicana de Mérida, Mérida
  - OCA Hospital, Monterrey N.L.
  - Hospital Central "Dr. Ignacio Morones Prieto", San Luis Potosi, SLP
  - Hospital "Dr. Angel Leaño", Zapopan, Jalisco
- Poland (7):
  - Swietokrzyskie Centrum Onkologii, Kielce
  - Wojewodzki Szpital Specjalistyczny im. L.Rydygiera, Krakow
  - Wojewodzki Szpital Specjalistyczny im. Mikolaja Kopernika, Regionalny Osrodek Onkologiczny, Lodz
  - Zaklad Opieki Zdrowotnej MSWiA z Warminsko-Mazurskim Centrum Onkologii, Olsztyn
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej, Opolskie Centrum Onkologii, Opole
  - Wielkopolskie Centrum Onkologii, Poznan
  - Centrum Onkologii Instytut im. M. Sklodowskiej-Curie, Warsaw
- Romania (2):
  - "Prof. Dr. I. Chiricuta" Institute of Oncology Medical Oncology and Radiotherapy II Department, Cluj-Napoca
  - Oradea Clinical County Hospital Department of Medical Oncology, Oradea
- Russia (14):
  - Regional Oncology Dispensary, Astrakhan
  - State Medical Institution Kursk Regional Oncology Dispensary Out-patient department, Kursk
  - Central Clinical Hospital #2 after MA Semashko OAO "RRW", Moscow
  - Moscow Scientific-Research Oncology Institute after P.A. Gertsen, Moscow
  - SI Russian Oncology Scientific Center after NN Blokhin RAMS, Moscow
  - PHI OAO RRW Railway Clinical Hospital at station Gorkiy, Nizhny Novgorod
  - Stavropol Regional Oncology Center, Pyatigorsk branch Out-patient department, Pyatigorsk
  - SIH Leningrad Regional Oncology Dispansery, Saint Petersburg
  - SPBSIH City Clinical Oncology Dispensary, Saint Petersburg
  - PHI Dorozhnaya Clinical Hospital at Saratov II Station of Pryvolzhskaya railway OAO Russian Railways, Saratov
  - Tambov Regional Oncological Dispensary Surgery Department, Tambov
  - Republican Clinical Oncological Dispenser Radiological Therapy, Ufa
  - State Medical Institution Regional Clinical Oncology Dispensary, Ulyanovsk
  - Sverdlovsk Regional Oncology Dispensary, Yekaterinburg
- Serbia (2):
  - Institute for Oncology and Radiology of Serbia, Belgrade
  - Military Medical Academy (MMA) Clinic for Maxillofacial Surgery, Belgrade
- Slovakia (5):
  - Teaching Hospital with Policlinic of F. D. Roosevelt Department of Otorhinolaryngology and Surgery, Banská Bystrica
  - Oncology Institute of St. Elisabeth Clinic of Stomatology and Maxillofacial Surgery, Bratislava
  - Teaching Hospital with Policlinic Bratislava 1st Clinic of Otorhinolaryngology, Bratislava
  - Vychodoslovensky oncologicky ustav a.s., Košice
  - Teaching Hospital with Policlinic Nové Zámky Clinic of Otorhinolaryngology, Nové Zámky
- Spain (6):
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital 12 de Octubre, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital Provincial de Pontevedra, Pontevedra
  - Hospital Universitario de Salamanca, Salamanca, Castilla Y León
- Ukraine (7):
  - Chernovtsy Regional Oncology Center, Chernivtsy
  - Kharkov Regional Clinical Oncology Dispensary, Kharkiv
  - Institute of Oncology of AMS of Ukraine, Kiev
  - Institute of Otolaryngology, Kiev
  - Volyn Regional Oncology Dispensary, Lutsk
  - Uzhgorod National University, Uzhhorod
  - Zaporozhye Regional Clinical Oncology Dispensary, Zaporizhzhya
- United Kingdom (3):
  - University Hospital Aintree, Liverpool
  - Royal Marsden Hospital, London
  - Christie Hospital, Manchester